CLINICAL TRIAL: NCT07166068
Title: The Effect of Mobilization With Movement Versus Sham Mobilization on Inflammatory Biomarkers in Patients With Knee Osteoarthritis.
Brief Title: The Effect of Mobilization on Inflammatory Biomarkers in Patients With Knee Osteoarthritis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jazan (Other Government)
Responsible Party: Principal Investigator, Abdulraouf Hamad Ayoub, Lecturer, Department of Physical Therapy, Principal Investigator, University of Jazan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: (HAPO-10-Z-001)
Record Dates: First submitted 2024-11-28; First posted 2025-09-10 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Knee Osteoarthritis
Keywords: Knee OA; MWM; Manual Therapy; CRP; ESR
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Musculoskeletal Manipulations; Movement; Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: While participants and outcome assessors are blinded to treatment allocation, therapists delivering the MWM and sham mobilization interventions are aware of the assigned treatment for each participant. However, therapists are blinded to all outcome measures, including pain scores, inflammatory marker results, and functional assessments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The intervention group will receive mobilization with movement for the affected knee with standard care (exercise program to strengthen the musculature of the knee).
  Interventions: Other: Manual Therapy (Mobilization with Movement); Other: Exercise
- Control Group (Placebo Comparator): The control group will receive sham mobilization with movement for the affected knee with standard care (exercise program to strengthen the musculature of the knee).
  Interventions: Other: Exercise; Other: sham mobilization

INTERVENTIONS:
Other: Manual Therapy (Mobilization with Movement) — A continuous glide to the tibia will be a combined simultaneously by whether medial, lateral, anterior, posterior, or rotational-during active knee flexion and extension repeated movement as applied by Mulligan.
  Arms: Intervention Group
Other: Exercise — standard care (exercise program to strengthen the musculature of the knee)
Other: sham mobilization — The therapist will simulate MWM by performing slight external rotation of the skin only. This mimics the tactile sensation of true MWM without affecting the underlying joint mechanics.
  Arms: Control Group

SUMMARY:
This study is designed to investigate whether a hands-on therapy called Mobilization with Movement (MWM) can reduce pain and inflammation in individuals with knee osteoarthritis (OA). The investigators will compare MWM to a sham treatment that resembles mobilization but does not involve the specific therapeutic movements. Both groups will also receive standard care, including exercise and education about managing knee OA.

A total of 40 adults (aged 18 years and older) with moderate to severe knee OA will be enrolled. Participants will be randomly assigned to either the MWM group or the sham group. Each intervention will be delivered twice per week over a four-week period.

Outcomes will include measures of inflammation obtained from blood samples, self-reported pain levels, and assessments of knee function before and after the intervention period. It is hypothesized that individuals allocated to the MWM group will demonstrate reduced inflammation and pain compared with those in the sham group. The findings of this study may help clarify the potential role of MWM as a treatment option for knee OA.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of unilateral or bilateral knee osteoarthritis (OA) according to the criteria of the American College of Rheumatology
* Age ≥ 18 years
* Kellgren-Lawrence grade 2 or 3 knee OA
* Pain intensity > 3 on a visual analogue scale (VAS)
* Body mass index (BMI) between 18.5 and 30 kg/m²

Exclusion Criteria:

* Knee or lower limb surgery within the last six months.
* Significant joint disorders (e.g., rheumatoid arthritis, gout, or other inflammatory arthritis).
* Recent significant acute infections.
* Contraindications to mobilization with movement.
* Current or recent use systemic glucocorticoids, intra-articular glucocorticoid injections or intra-articular hyaluronic acid injections.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2026-02-20 (Estimated); Study Completion 2026-04-20 (Estimated)

PRIMARY OUTCOMES:
C-Reactive Protein (CRP) | Baseline and 4 weeks post-intervention.
  CRP levels will be measured in unit of measure (mg/L) using a high-sensitivity assay.
Erythrocyte Sedimentation Rate (ESR) | Baseline and 4 weeks post-intervention.
  ESR will be measured in mm/hr using the Westergren method.

SECONDARY OUTCOMES:
Pain Intensity | The outcome measure will be assessed at the baseline and 4 weeks post-intervention.
  The pain intensity will be assessed using a Visual Analog Scale (VAS) ranging from 0 (no pain) to 10 (worst pain imaginable).
Functional Status | The outcome measure will be assessed at the baseline and 4 weeks post-intervention.
  Functional status will be evaluated using the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) function subscale.

CONTACTS AND LOCATIONS:
Locations (1):
- Jazan University Hospital, Jizan, Jazan Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Li LL, Hu XJ, Di YH, Jiao W. Effectiveness of Maitland and Mulligan mobilization methods for adults with knee osteoarthritis: A systematic review and meta-analysis. World J Clin Cases. 2022 Jan 21;10(3):954-965. doi: 10.12998/wjcc.v10.i3.954. PMID 35127909
- [Background] Shabbir M, Gul I, Asghar E, Muhammad N, Mehjabeen H, Rafiq I, Arshad N. Effectiveness Of Maitland's Mobilization And Conventional Physical Therapy On Synovial Biomarkers In Patients With Knee Osteoarthritis; A Randomized Control Trial. Webology. 2022 Apr 1;19(2)
- [Background] Hanada M, Takahashi M, Furuhashi H, Koyama H, Matsuyama Y. Elevated erythrocyte sedimentation rate and high-sensitivity C-reactive protein in osteoarthritis of the knee: relationship with clinical findings and radiographic severity. Ann Clin Biochem. 2016 Sep;53(Pt 5):548-53. doi: 10.1177/0004563215610142. Epub 2015 Sep 17. PMID 26384360
- [Background] Zaki NA, Saleem TH, Said E, Hassan MH. Evidence of contributory role of inflammation in patients with knee osteoarthritis. SVU-International Journal of Medical Sciences. 2020 Jan 1;3(1):1-6.
- [Background] Althomali OW, Amin J, Acar T, Shahanawaz S, Talal Abdulrahman A, Alnagar DK, Almeshari M, Alzamil Y, Althomali K, Alshoweir N, Althomali O, Aldhahi MI, Bin Sheeha BH. Prevalence of Symptomatic Knee Osteoarthritis in Saudi Arabia and Associated Modifiable and Non-Modifiable Risk Factors: A Population-Based Cross-Sectional Study. Healthcare (Basel). 2023 Mar 2;11(5):728. doi: 10.3390/healthcare11050728. PMID 36900733
- [Background] Cui A, Li H, Wang D, Zhong J, Chen Y, Lu H. Global, regional prevalence, incidence and risk factors of knee osteoarthritis in population-based studies. EClinicalMedicine. 2020 Nov 26;29-30:100587. doi: 10.1016/j.eclinm.2020.100587. eCollection 2020 Dec. PMID 34505846
- See also: OARSI is the premier international organization for scientists and healthcare professionals focused on osteoarthritis research, prevention, and treatment. — https://oarsi.org/